CLINICAL TRIAL: NCT01151800
Title: Using Interactive Voice Response To Improve Disease Management and Compliance With Acute Coronary Syndrome Best Practice Guidelines
Brief Title: Using Automated Calls To Improve Compliance With Acute Coronary Syndrome Best Practice Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: The Change Foundation (Other)
Responsible Party: Heather Sherrard, VP Clinical Services, University of Ottawa Heart Institute
Allocation: Randomized | Purpose: Treatment
Other Study IDs: UOHI 2006-128
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Acute Coronary Syndrome; Medication Adherence
Keywords: ACS; Interactive Voice Response Technology; Best Practice Guidelines; Health Care Utilization; Outcome Assessment
MeSH Terms: conditions — Acute Coronary Syndrome; Medication Adherence; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVR group (Experimental)
  Interventions: Other: Using IVR to maintain ACS patients on best practice guidelines
- Usual care (No Intervention)

INTERVENTIONS:
Other: Using IVR to maintain ACS patients on best practice guidelines
  Arms: IVR group

SUMMARY:
The purpose of this study is to determine whether interactive voice response (IVR) technology can be used to bring post discharge care for acute coronary syndrome (ACS) closer to best practice guidelines (BPGs).

The study hypothesis is that ACS patients who are contacted by IVR technology will be more likely to receive care as recommended in the BPGs than those followed by usual care.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is a significant public-health problem in Canada and worldwide with 20,000 Canadians dying of myocardial infarction and 42,000 dying of coronary artery disease in 1999. Large clinical trials have provided evidence for the development of standardized best practice guidelines (BPG) and compliance with these guidelines have significantly improved survival. Despite the development and dissemination of BPG, their application in patients with ACS is suboptimal. This randomized control trial will use 2 groups: IVR and usual care. Patients in the IVR group will receive 5 automated calls at 1,3,6,9 and 12 months consisting of predetermined questions related to medication management, smoking cessation, diet, exercise and education as recommended by the ACC/AHA BPG for ACS. Responses are captured in a database allowing for interventions to maintain patients on BPG as needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged from the UOHI with ACS (acute myocardial infarction, STEMI or NSTEMI)
* Patients who have a land line telephone service at home
* Patients who speak English or French

Exclusion Criteria:

* Patients discharged to a care facility or transferred to another health care institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1608 (Actual)
Dates: Start 2006-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Compliance with BPGs | 1 year

SECONDARY OUTCOMES:
Utilization of health care resources: emergency visits, unscheduled physician visits and hospitalization and patient satisfaction | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada